CLINICAL TRIAL: NCT05996601
Title: Evaluation of Selected Improved Outcomes Among Patients With Diabetes and/or Hypertension in Designated Community Pharmacies in a Metropolitan City - An Intervention Study
Brief Title: Evaluation of Improved Outcomes Among Ambulatory Diabetes and/or Hypertensive Patients - an Intervention Study (CPCLINT)
Acronym: CPCLINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Akinniyi Akinbiyi Aje, Experiential Training Coordinator and Sub-Dean Undergraduate (Integrated), University of Ibadan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CPINTCLI
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Diabetes; Hypertension; Interventional study; Health literacy; Physical activity; Medication adherence; Pharmacist; Community pharmacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus; Motor Activity; Medication Adherence | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): All participants would undergo educational intervention by pharmacist.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — Educational materials would be given to all the participants. They would also be followed up by pharmacist.

SUMMARY:
The goal of this interventional study is to compare improved outcomes among diabetes and/or hypertensive patients sequel to educational intervention. The study aims to answer the following questions:

* What are the patients' levels of health literacy, medication adherence, disease knowledge, attitude to disease, physical activity?
* Does educational intervention by pharmacists improve health outcomes of patients with diabetes and/or hypertension?
* Are there associations between patient-related variables such as health literacy, medication adherence, disease knowledge, attitude to disease? Participants' anthropometric measurements and point-of-care testing for disease monitoring e.g., blood pressure, blood glucose would be carried out. Baseline assessment of participants would be done to evaluate their levels of health literacy, medication adherence, disease knowledge, attitude to disease, physical activity.

Patients' baseline assessment would be carried out, after which they would receive educational materials and would be followed up by pharmacist. The baseline assessments would be repeated at three and six months after the intervention to measure the effectiveness of the intervention.

DETAILED DESCRIPTION:
The anthropometric measurements would include weight, height, waist circumference, hip circumference, from which the body mass index and waist-hip ration would be calculated.

The assessment of the disease knowledge and attitude would be done using validated semi-structured questionnaires earlier designed by the principal investigator and used among ambulatory patients with diabetes and/or hypertension accessing care in tertiary healthcare facilities. The validated International Physical Activity Questionnaire (IPAQ) would be utilized for participants' physical activity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 18 years of age
* Patients must be diagnosed with diabetes and/or hypertension
* Patients must be on at least one medication
* Patients who access one of the selected community pharmacies for prescription refill

Exclusion Criteria:

* Non-consented patients
* Patients not based at the study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | 6 months
  Participants' blood pressure in mmHg measured at baseline, 3- and 6-month postintervention would be compared to find out if there are changes.
Blood glucose control of participants | 6 months
  Fasting blood glucose in mg/dL measured at baseline, 3- and 6-month postintervention. would be compared.
Participants' level of disease knowledge and attitude | 6 months
  The knowledge and attitude scale in the semi-structured questionnaire would be evaluated at baseline, 3- and 6-month postintervention.
Participants' body mass index calculated by dividing weight in kilograms by the square of height in meters. | 6 months
  Participants weight in kilograms and height in meters would be measured at baseline, 3- and 6-month postintervention. Their body mass index would be compared to find out if there are changes.
Medication adherence of participants using a 4-item medication adherence scale | 6 months
  Participants' medication adherence would be evaluated at baseline, 3- and 6-month postintervention using Morisky, Green and Levine 4-item medication adherence scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aduke E Ipingbemi, PhD, Study Director — University of Ibadan, Nigeria.
Locations (1):
- Department of Clinical Pharmacy and Pharmacy Administration, Faculty of Pharmacy, University of Ibadan., Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No
I might not share this based on sensitive nature of data to be collected. However, the group data generated would be shared through publications in peer-reviewed journals for public consumption.

REFERENCES:
- [Background] Adeloye D, Owolabi EO, Ojji DB, Auta A, Dewan MT, Olanrewaju TO, Ogah OS, Omoyele C, Ezeigwe N, Mpazanje RG, Gadanya MA, Agogo E, Alemu W, Adebiyi AO, Harhay MO. Prevalence, awareness, treatment, and control of hypertension in Nigeria in 1995 and 2020: A systematic analysis of current evidence. J Clin Hypertens (Greenwich). 2021 May;23(5):963-977. doi: 10.1111/jch.14220. Epub 2021 Feb 18. PMID 33600078
- [Background] Uloko AE, Musa BM, Ramalan MA, Gezawa ID, Puepet FH, Uloko AT, Borodo MM, Sada KB. Prevalence and Risk Factors for Diabetes Mellitus in Nigeria: A Systematic Review and Meta-Analysis. Diabetes Ther. 2018 Jun;9(3):1307-1316. doi: 10.1007/s13300-018-0441-1. Epub 2018 May 14. PMID 29761289
- [Background] Milosavljevic A, Aspden T, Harrison J. Community pharmacist-led interventions and their impact on patients' medication adherence and other health outcomes: a systematic review. Int J Pharm Pract. 2018 Oct;26(5):387-397. doi: 10.1111/ijpp.12462. Epub 2018 Jun 21. PMID 29927005
- [Background] Rajiah K, Sivarasa S, Maharajan MK. Impact of Pharmacists' Interventions and Patients' Decision on Health Outcomes in Terms of Medication Adherence and Quality Use of Medicines among Patients Attending Community Pharmacies: A Systematic Review. Int J Environ Res Public Health. 2021 Apr 21;18(9):4392. doi: 10.3390/ijerph18094392. PMID 33918990